CLINICAL TRIAL: NCT01228617
Title: Single-dose Pharmacokinetics of Oral Nicotine Replacement Products - An Exploratory Study in Healthy Volunteers
Brief Title: Single-dose Pharmacokinetics of Oral Nicotine Replacement Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A6431114-NICTDP1063
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- A1 Short, no buffer (Experimental): Nicotine / not yet marketed
  Interventions: Drug: Nicotine
- A2 Short, low buffer (Experimental): Nicotine / not yet marketed
  Interventions: Drug: Nicotine
- A3 Short, high buffer (Experimental): Nicotine / not yet marketed
  Interventions: Drug: Nicotine
- B1 Long, no buffer (Experimental): Nicotine / not yet marketed
  Interventions: Drug: Nicotine
- B2 Long, low buffer (Experimental): Nicotine / not yet marketed
  Interventions: Drug: Nicotine
- B3 Long, high buffer (Experimental): Nicotine / not yet marketed
  Interventions: Drug: Nicotine
- R = Nicotine Gum (Active Comparator): Nicorette® Gum
  Interventions: Drug: Nicotine Gum

INTERVENTIONS:
Drug: Nicotine — Following a 12-hour nicotine abstinence period, subjects receive a single 2 mg dose of their assigned nicotine replacement therapy in the morning of the treatment visit day
  Other Names: Not yet marketed
  Arms: A1 Short, no buffer; A2 Short, low buffer; A3 Short, high buffer; B1 Long, no buffer; B2 Long, low buffer; B3 Long, high buffer
Drug: Nicotine Gum — Following a 12-hour nicotine abstinence period, subjects will be instructed to chew the gum once every 2 seconds, for 30 minutes.
  Other Names: Nicorette®
  Arms: R = Nicotine Gum

SUMMARY:
This is an explorative study comparing new prototypes of Nicotine Replacement Products with Nicorette® gum.

DETAILED DESCRIPTION:
This study included 40 subjects who were randomly assigned to one of eight treatment sequences. In four of the sequences, the three prototypes with the shorter dissolution time and the reference were used; in the remaining four sequences, the three prototypes with the longer dissolution time and the reference were used. Hence, half of the subjects received the Short prototypes and half received the Long prototypes. Subjects in both treatment groups (short and long) attended four treatment visits, each of 11 hours' duration, and periods of at least 36 hours' duration between treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers, smoking at least 10 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration | Baseline to 10 hours post-dose
  The maximum observed nicotine concentration in plasma (Cmax)
Area under the Curve | 10 hours post-dose
  The area under the plasma concentration-vs.-time curve until the last measurable concentration (AUCt)and the area under the plasma concentration-vs.-time curve until infinity (AUC∞)

SECONDARY OUTCOMES:
Time to Maximum Concentration | 10 hours post-dose
  Time to Maximum Concentration (Tmax)
Residual Nicotine | 30 minutes
  The amount of residual nicotine in the product after being chewed.
Dissolution Time | 10 hours post-dose
  Actual time required for oral dissolution of new NRT products following product administration

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Clinical Trial Unit, Clinical Research and Trial Centre, Lund, Sweden